CLINICAL TRIAL: NCT06148701
Title: The Preoperative Anesthesia automatiC systeM for triAge and screeNing (PACMAN) as a Model for Recognition of Patients Who May Screened by Phone: a Retrospective Cohort Study
Brief Title: Preoperative Anesthesia Automatic System:a Retrospective Cohort Study
Acronym: PACMAN
Status: Completed | Type: Observational
Sponsor: Jeroen Bosch Ziekenhuis (Other)
Responsible Party: Sponsor
Other Study IDs: 2021.08.06.01
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Surgical Procedure, Unspecified; Anesthesia; Assessment
Keywords: Anaesthetists / Health Care Surveys / Preoperative Care / Triage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate of PACMAN triage system is able to discern patient who may be safely screened by phone

DETAILED DESCRIPTION:
PACMAN triage system consists of a health questionnaire and an algorithm. Patient were called up by registered nurses and asked to answer the questionnaire. Patients answers were applied to PACMAN algorithm to determine what kind of screening patient should receive: in person or by phone.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old, scheduled for elective clinical interventions under procedural sedation and all types of elective medium or low risk surgery with anaesthetic guidance, as defined by the European Society of Anaesthesia (ESA) guidelines.

Exclusion Criteria:

* <18 years. Patients scheduled for emergency and high-risk surgery were excluded as the policy of our department dictates that these patients must always be seen in person, according to ESA guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for all kind of surgical procedures except cardiac surgery and intracranial surgery
Sampling Method: Non-Probability Sample
Enrollment: 1019 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Reduction of the number of in person consultations | between start inclusion and 6 months after start inclusion
  In 2019 all patients were screened in person. Aim of the study is to evaluate whether implementation of PACMAN leads to a significant reduction of the number of in person consultations

SECONDARY OUTCOMES:
Reliability of PACMAN | between start inclusion and 6 months after start inclusion
  Reliability of the triage procedure was evaluated by verifying the PACMAN outcome (PhC vs in-PC) against the assigned ASA-PS classification. Patients scheduled for a PhC were considered to be accurately triaged if classified ASA-PS I-II or III with stable comorbidities. Patients scheduled for an in-PC were considered to be accurately triaged if classified ASA-PS III with unstable comorbidities or IV.
Patients outcome | between start inclusion and 6 months after start inclusion
  To measure the impact of PACMAN on patient outcomes we evaluated the occurrence of perioperative unanticipated adverse events (UAE). An anaesthesia-related UAE was defined as an event causing mortality or morbidity, occurring during the perioperative period or up to seven days after surgery and requiring special medical treatment or prolongation of hospitalisation beyond the expected length of stay. Data concerning perioperative UAE were collected by reviewing the EMR of patients who had undergone surgery.
Cost-effectiveness | between start inclusion and 6 months after start inclusion
  we examined cost-effectiveness and efficiency by determining the time taken by screening staff for a single PhC or in-PC and the average number of patients screened before and after implementation of PACMAN along with related staff costs.

CONTACTS AND LOCATIONS:
Overall Officials: Barbe Pieters, Dr.PhD, Principal Investigator — Jeroen Bosch Hospital, 's Hertogenbosch The Netherlands
Locations (1):
- Jeroen Bosch Ziekenhuis, 's-Hertogenbosch, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Di Biase M, van der Zwaard B, Aarts F, Pieters B. Pre-operative triAge proCedure to streaMline elective surgicAl patieNts (PACMAN) improves efficiency by selecting patients eligible for phone consultation: A retrospective cohort study. Eur J Anaesthesiol. 2024 Nov 1;41(11):813-820. doi: 10.1097/EJA.0000000000002055. Epub 2024 Sep 9. PMID 39252617